CLINICAL TRIAL: NCT05829655
Title: Measuring Acute Drug Demand in Humans
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00344798; R01DA055634 (NIH)
Record Dates: First submitted 2023-04-13; First posted 2023-04-26 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder; Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Suvorexant (20mg/day) (Experimental): Double blind administration of suvorexant once per day during residential stay until discharge
  Interventions: Drug: Drug A (Blinded Drug); Drug: Drug B (Blinded Drug); Drug: Drug C (Blinded Drug); Drug: Drug D (Blinded Drug); Drug: Suvorexant (20mg/day)
- Placebo (Placebo Comparator): Double blind administration of placebo once per day during residential stay until discharge
  Interventions: Drug: Drug A (Blinded Drug); Drug: Drug B (Blinded Drug); Drug: Drug C (Blinded Drug); Drug: Drug D (Blinded Drug); Drug: Placebo

INTERVENTIONS:
Drug: Drug A (Blinded Drug) — Participants will receive a double-blinded oral study medication as part of their daily sessions and will provide feedback regarding the effects of the medication on various measures. Though the study medications are FDA approved, they are being used here for a non-FDA approved purpose (though the FDA has provided permission to use these drugs in this study).
Drug: Drug B (Blinded Drug) — Participants will receive a double-blinded oral study medication as part of their daily sessions and will provide feedback regarding the effects of the medication on various measures. Though the study medications are FDA approved, they are being used here for a non-FDA approved purpose (though the FDA has provided permission to use these drugs in this study).
Drug: Drug C (Blinded Drug) — Participants will receive a double-blinded oral study medication as part of their daily sessions and will provide feedback regarding the effects of the medication on various measures. Though the study medications are FDA approved, they are being used here for a non-FDA approved purpose (though the FDA has provided permission to use these drugs in this study).
Drug: Drug D (Blinded Drug) — Participants will receive a double-blinded oral study medication as part of their daily sessions and will provide feedback regarding the effects of the medication on various measures. Though the study medications are FDA approved, they are being used here for a non-FDA approved purpose (though the FDA has provided permission to use these drugs in this study).
Drug: Suvorexant (20mg/day) — Double blind administration of suvorexant once per day during residential stay until discharge.
  Arms: Suvorexant (20mg/day)
Drug: Placebo — Double blind administration of placebo once per day during residential stay until discharge.
  Arms: Placebo

SUMMARY:
This research is being done to evaluate whether suvorexant may reduce the use of, subjective liking, and demand for various drugs.

DETAILED DESCRIPTION:
This research is being done to evaluate whether suvorexant may reduce the use of, subjective liking, and demand for various drugs. Suvorexant is not approved as a treatment to reduce drug use but is approved by the Food and Drug Administration (FDA) to treat insomnia (trouble falling asleep or staying asleep). This study consists of a screening visit and an approximate 14 to 16 day inpatient (overnight) stay at the Johns Hopkins Bayview Medical Center. Participants will be stabilized on hydromorphone, randomly assigned to receive either suvorexant or placebo, and complete 5 experimental sessions that include taking blinded study medications.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old
* Meets Diagnostic and Statistical Manual-5 criteria for Opioid Use Disorder (OUD) (moderate or severe)
* Lifetime substance use history criterion [blinded]
* Medically cleared to take suvorexant and blinded study medications
* Be in good general health based on a physical examination, medical history, vital signs, and screening urine and blood tests

Exclusion Criteria:

* Pregnant or breast feeding
* Seeking opioid use treatment
* Significant mental health or physical disorder that is expected to interfere with study participation as assessed by the study physicians or medical staff
* Known contraindications or allergies to suvorexant and/or the blinded study medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Demand Intensity | Upon completion of experimental session (~8 hours post drug administration)
  Consumption of blinded drug at unconstrained price as measured by an incentivized demand task. Minimum value is 0, maximum value is not constrained. Higher scores indicate more drug consumption at unconstrained price (a worse outcome).
Demand Elasticity | Upon completion of experimental session (~8 hours post drug administration)
  Changes in blinded drug consumption with changes in price as measured by an incentivized demand task. There is no minimum or maximum value. Higher scores indicate greater drug price sensitivity (a better outcome).
Cross-Price Elasticity | After Experimental Session 4
  Change in consumption of price-fixed good based on change in price of price varying good. Positive values indicate a substitute, negative values indicate a complement, and zero values indicate an independent commodity.

SECONDARY OUTCOMES:
Total Mean Sleep Time | Through study completion, up to two weeks
  Mean total number of minutes slept per night as measured by actigraphy and self-reported sleep diary. Mean total sleep time will be collected daily.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Strickland, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States